CLINICAL TRIAL: NCT00366548
Title: A Phase 3, Randomized, Double-blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine Manufactured With and Without Polysorbate 80 in Healthy Infants Given in a 2-, 3-, 4-, and 12-Month Schedule With Routine Pediatric Vaccinations
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6096A1-009
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-07

CONDITIONS: Vaccines, Pneumococcal
Keywords: Vaccine; Infant
MeSH Terms: interventions — Polysorbates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine with Polysorbate 80
- 2 (Active Comparator)
  Interventions: Biological: 13 valent pneumococcal conjugate vaccine without Polysorbate 80

INTERVENTIONS:
Biological: 13 valent pneumococcal conjugate vaccine with Polysorbate 80
  Arms: 1
Biological: 13 valent pneumococcal conjugate vaccine without Polysorbate 80
  Arms: 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine manufactured with Polysorbate 80 compared to a 13-valent pneumococcal conjugate (13vPnC) manufactured without Polysorbate 80 when given concomitantly with routine paediatric vaccinations.

ELIGIBILITY:
Inclusion criteria:

1. Aged 2 months (42 through 98 days) at the time of enrollment.
2. Available for the entire study period and whose parent(s)/legal guardian(s) could be reached by telephone.
3. In good health as determined by medical history, physical examination, and judgment of the investigator.
4. Parent(s)/legal guardian(s) were able to complete all relevant study procedures during study participation.

Exclusion criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. Previous vaccination with Hib conjugate, diphtheria, tetanus, pertussis, or polio vaccines.
3. A previous anaphylactic reaction to any vaccine or vaccine-related component.
4. Contraindication to vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, hepatitis B, or pneumococcal vaccines.
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
6. Known or suspected immune deficiency or suppression.
7. History of culture-proven invasive disease caused by S pneumoniae.
8. Major known congenital malformation or serious chronic disorder.
9. Significant neurological disorder or history of seizure (including febrile seizure), or significant stable or evolving disorders (such as cerebral palsy, encephalopathy, or hydrocephalus), or other significant disorders. This did not include resolving syndromes because of birth trauma such as Erb palsy.
10. Receipt of blood products or γ-globulin (including hepatitis B immunoglobulin and monoclonal antibodies [eg, Synagis]).

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com
Locations (11):
- Poland (11):
  - Bydgoszcz
  - Dębica
  - Krakow
  - Lodz
  - Lubartów
  - Lublin
  - Oborniki Śląskie
  - Poznan
  - Siemianowice Śląskie
  - Torun
  - Trzebnica

REFERENCES:
- [Derived] Gadzinowski J, Tansey SP, Wysocki J, Kopinska E, Majda-Stanislawska E, Czajka H, Korbal P, Pietrzyk JJ, Baker SA, Giardina PC, Gruber WC, Emini EA, Scott DA. Safety and immunogenicity of a 13-valent pneumococcal conjugate vaccine manufactured with and without polysorbate 80 given to healthy infants at 2, 3, 4 and 12 months of age. Pediatr Infect Dis J. 2015 Feb;34(2):180-5. doi: 10.1097/INF.0000000000000511. PMID 25126854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Poland from November 2006 to December 2006.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC With (+) Polysorbate 80: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) with (+) P80 coadministered with combination vaccine containing diphtheria, tetanus, acellular pertussis, inactivated poliovirus, and conjugated Hib antigens (Pentaxim) and hepatitis B recombinant vaccine adsorbed (Engerix-B) at approximately 2 months of age, Pentaxim at approximately 3 months and 4 months of age (infant series), and combined vaccine containing attenuated measles, mumps, and rubella viruses (Priorix) at 12 months of age (toddler dose).
- 13vPnC Without (-) Polysorbate 80: Participants received one single 0.5mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) without (-) P80 coadministered with combination vaccine containing diphtheria, tetanus, acellular pertussis, inactivated poliovirus, and conjugated Hib antigens (Pentaxim) and hepatitis B recombinant vaccine adsorbed (Engerix-B) at approximately 2 months of age, Pentaxim at approximately 3 months and 4 months of age (infant series), and combined vaccine containing attenuated measles, mumps, and rubella viruses (Priorix) at 12 months of age (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC With (+) Polysorbate 80 | 13vPnC Without (-) Polysorbate 80
Started | 250 | 250
Vaccinated Dose 1 | 250 | 250
Vaccinated Dose 2 | 246 | 249
Vaccinated Dose 3 | 246 | 247
Completed | 246 | 245
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1
Period: After Infant Series
Arm/Group | 13vPnC With (+) Polysorbate 80 | 13vPnC Without (-) Polysorbate 80
Started | 246 | 245
Completed | 240 | 244
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC With (+) Polysorbate 80 | 13vPnC Without (-) Polysorbate 80
Started | 240 | 244
Completed | 240 | 244
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC With (+) Polysorbate 80 | 13vPnC Without (-) Polysorbate 80 | Total
Number analyzed (Participants) | 250 | 250 | 500
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.5) | 2.1 (0.5) | 2.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 122 | 244
  Male | 128 | 128 | 256

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Antibody Level ≥0.35μg/mL in 13vPnC+P80 Group Relative to 13vPnC-80 Group After the Infant Series
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (at 5 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations, (n) = number of participants with a determinate immunoglobulin G (IgG) antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC + Polysorbate 80 After the Infant Series: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
- 13vPnC - Polysorbate 80 After the Infant Series: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
Arm/Group | 13vPnC + Polysorbate 80 After the Infant Series | 13vPnC - Polysorbate 80 After the Infant Series
Number analyzed (Participants) | 238 | 238
percentage of participants
  Common Serotypes - Serotype 4 (n=222,224) | 93.3 [89.3 to 96.1] | 94.1 [90.3 to 96.7]
  Common Serotypes - Serotype 6B (n=145,158) | 60.9 [54.4 to 67.2] | 66.4 [60.0 to 72.4]
  Common Serotypes - Serotype 9V (n=231,232) | 97.1 [94.0 to 98.8] | 97.5 [94.6 to 99.1]
  Common Serotypes - Serotype 14 (n=225,232) | 94.5 [90.8 to 97.1] | 97.5 [94.6 to 99.1]
  Common Serotypes - Serotype 18C (n=233,233) | 97.9 [95.2 to 99.3] | 97.9 [95.2 to 99.3]
  Common Serotypes - Serotype 19F (n=228,234) | 95.8 [92.4 to 98.0] | 98.3 [95.8 to 99.5]
  Common Serotypes - Serotype 23F (n=205,220) | 86.1 [81.1 to 90.3] | 92.4 [88.3 to 95.5]
  Additional Serotypes - Serotype 1 (n=228,220) | 95.8 [92.4 to 98.0] | 92.4 [88.3 to 95.5]
  Additional Serotypes - Serotype 3 (n=233,236) | 97.9 [95.2 to 99.3] | 99.2 [97.0 to 99.9]
  Additional Serotypes - Serotype 5 (n=224,220) | 94.1 [90.3 to 96.7] | 92.4 [88.3 to 95.5]
  Additional Serotypes - Serotype 6A (n=206,205) | 86.6 [81.6 to 90.6] | 86.1 [81.1 to 90.3]
  Additional Serotypes - Serotype 7F (n=235,237) | 98.7 [96.4 to 99.7] | 99.6 [97.7 to 100.0]
  Additional Serotypes - Serotype 19A (n=235,238) | 98.7 [96.4 to 99.7] | 100.0 [98.5 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lowest limit of the 2-sided 95% CI for the difference between the 2 groups > -10%; Difference = -0.8, 95% CI [-5.4 to 3.7]
Statistical Analysis 2: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -5.5, 95% CI [-14.2 to 3.3]
Statistical Analysis 3: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.4, 95% CI [-3.7 to 2.8]
Statistical Analysis 4: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.9, 95% CI [-6.9 to 0.7]
Statistical Analysis 5: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-3.0 to 3.0]
Statistical Analysis 6: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -2.5, 95% CI [-6.1 to 0.6]
Statistical Analysis 7: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -6.3, 95% CI [-12.1 to -0.7]
Statistical Analysis 8: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 1 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 3.4, 95% CI [-0.9 to 7.9]
Statistical Analysis 9: Comparison: 13vPnC - Polysorbate 80 After the Infant Series; For serotype 3 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.3, 95% CI [-4.1 to 1.1]
Statistical Analysis 10: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 5 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 1.7, 95% CI [-3.0 to 6.4]
Statistical Analysis 11: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 6A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-5.8 to 6.7]
Statistical Analysis 12: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 7F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.8, 95% CI [-3.2 to 1.2]
Statistical Analysis 13: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 19A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.3, 95% CI [-3.6 to 0.3]

2. Secondary Outcome: Percentage of Participants Achieving Antibody Level ≥ 0.35 μg/mL in the 13vPnC Group After the Toddler Dose
Description: Percentages of participants achieving World Health Organization (WHO) predefined antibody threshold ≥ 0.35 μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after the toddler dose (at 13 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations, (n) = number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 13vPnC + Polysorbate 80 After Toddler Dose: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at approximately 2 months of age, Pentaxim at approximately 3 months and 4 months of age (infant doses), and Priorix at 12 months of age (toddler dose).
- 13vPnC - Polysorbate 80 After Toddler Dose: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at the 2 month visit, Pentaxim at the 3 and 4 month visits, and Priorix at 12 months of age (toddler dose).
Arm/Group | 13vPnC + Polysorbate 80 After Toddler Dose | 13vPnC - Polysorbate 80 After Toddler Dose
Number analyzed (Participants) | 227 | 238
percentage of participants
  Common Serotypes - Serotype 4 (n=226,238) | 99.6 [97.6 to 100.0] | 99.6 [97.7 to 100.0]
  Common Serotypes - Serotype 6B (n=225,237) | 99.6 [97.5 to 100.0] | 99.2 [97.0 to 99.9]
  Common Serotypes - Serotype 9V (n=226,238) | 99.6 [97.6 to 100.0] | 100.0 [98.5 to 100.0]
  Common Serotypes - Serotype 14 (n=226,238) | 99.6 [97.6 to 100.0] | 99.6 [97.7 to 100.0]
  Common Serotypes - Serotype 18C (n=226,238) | 100.0 [98.4 to 100.0] | 99.6 [97.7 to 100.0]
  Common Serotypes - Serotype 19F (n=226,237) | 99.1 [96.8 to 99.9] | 98.7 [96.3 to 99.7]
  Common Serotypes - Serotype 23F (n=226,238) | 98.7 [96.2 to 99.7] | 99.6 [97.7 to 100.0]
  Additional Serotypes - Serotype 1 (n=226,238) | 100.0 [98.4 to 100.0] | 99.2 [97.0 to 99.9]
  Additional Serotypes - Serotype 3 (n=223,236) | 95.1 [91.3 to 97.5] | 94.5 [90.8 to 97.0]
  Additional Serotypes - Serotype 5 (n=226,238) | 99.6 [97.6 to 100.0] | 100.0 [98.5 to 100.0]
  Additional Serotypes - Serotype 6A (n=226,237) | 99.6 [97.6 to 100.0] | 100.0 [98.5 to 100.0]
  Additional Serotypes - Serotype 7F (n=226,238) | 100.0 [98.4 to 100.0] | 100.0 [98.5 to 100.0]
  Additional Serotypes - Serotype 19A (n=226,238) | 100.0 [98.4 to 100.0] | 100.0 [98.5 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 4 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.0, 95% CI [-2.1 to 1.9]
Statistical Analysis 2: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 6B the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-1.7 to 2.6]
Statistical Analysis 3: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 9V the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.4, 95% CI [-2.4 to 1.1]
Statistical Analysis 4: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 14 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.0, 95% CI [-2.1 to 1.9]
Statistical Analysis 5: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 18C the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-1.2 to 2.3]
Statistical Analysis 6: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 19F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.4, 95% CI [-2.0 to 2.9]
Statistical Analysis 7: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 23F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.9, 95% CI [-3.4 to 1.1]
Statistical Analysis 8: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 1 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.8, 95% CI [-0.8 to 3.0]
Statistical Analysis 9: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 3 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.6, 95% CI [-3.7 to 4.9]
Statistical Analysis 10: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 5 the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.4, 95% CI [-2.4 to 1.1]
Statistical Analysis 11: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 6A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -0.4, 95% CI [-2.4 to 1.2]
Statistical Analysis 12: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 7F the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 1.6]
Statistical Analysis 13: Comparison: 13vPnC + Polysorbate 80 After Toddler Dose vs 13vPnC - Polysorbate 80 After Toddler Dose; For serotype 19A the difference in percentages between the two groups (13vPnC - 7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-1.7 to 1.6]

3. Other Pre Specified Outcome: Percent of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were collected using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (Sig) (present and interfered with limb movement). Swelling and redness were scaled as Any (swelling or redness present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (Mod) (2.5 to 7.0 cm); Severe (>7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4-days after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC + P80 Dose 1 Infant Series: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age(infant series, Dose 1).
- 13vPnC - P 80 Dose 1 Infant Series: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age (infant series, Dose 1).
- 13vPnC + P80 Dose 2 Infant Series: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 months age (infant series, Dose 2).
- 13vPnC - P80 Dose 2 Infant Series: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 months age (infant series, Dose 2).
- 13vPnC + P80 Dose 3 Infant Series: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant series, Dose 3).
- 13vPnC - P80 Dose 3 Infant Series: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant series, Dose 3).
- 13vPnC + P80 Toddler Dose: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant series), and Priorix at 12 months of age (toddler dose).
- 13vPnC - P80 Toddler Dose: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant series), and Priorix at 12 months of age (toddler dose).
Arm/Group | 13vPnC + P80 Dose 1 Infant Series | 13vPnC - P 80 Dose 1 Infant Series | 13vPnC + P80 Dose 2 Infant Series | 13vPnC - P80 Dose 2 Infant Series | 13vPnC + P80 Dose 3 Infant Series | 13vPnC - P80 Dose 3 Infant Series | 13vPnC + P80 Toddler Dose | 13vPnC - P80 Toddler Dose
Number analyzed (Participants) | 250 | 250 | 246 | 249 | 246 | 247 | 240 | 244
Percentage of Participants
  Tenderness-Any (n=238,237,228,229,210,216,178,188) | 27.7 | 32.9 | 26.8 | 32.8 | 24.8 | 23.1 | 42.1 | 43.1
  Tenderness-Sig (n=235,233,220,221,203,211,160,165) | 2.1 | 4.3 | 0.9 | 0.5 | 1.5 | 1.9 | 2.5 | 1.2
  Swelling-Any (n=236,239,228,228,210,225,174,181) | 22.9 | 30.5 | 25.0 | 36.4 | 36.7 | 38.2 | 29.9 | 34.8
  Swelling-Mild (n=236,236,227,226,209,221,169,178) | 18.2 | 24.2 | 20.3 | 31.9 | 32.5 | 33.5 | 26.6 | 29.8
  Swelling-Mod (n=236,236,224,224,208,217,164,171) | 11.9 | 14.4 | 11.2 | 14.3 | 13.9 | 17.5 | 12.2 | 19.9
  Swelling-Severe(n=235,233,220,221,203,211,159,164) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=238,238,232,231,216,226,178,200) | 29.8 | 39.5 | 38.8 | 48.5 | 46.8 | 50.0 | 42.1 | 52.0
  Redness-Mild (n=238,235,232,230,215,226,176,194) | 28.2 | 35.7 | 38.4 | 47.0 | 46.5 | 46.9 | 35.8 | 46.4
  Redness-Mod (n=235,232,220,222,206,211,164,173) | 2.1 | 4.3 | 1.4 | 3.2 | 3.9 | 9.0 | 12.8 | 19.7
  Redness-Severe (n=235,231,220,221,203,211,159,164) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.6

4. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever [Fv] ≥ 37.5 degrees Celsius [C], fever ≥ 38 C but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased (decr)appetite, irritability, increased (incr)sleep, decreased sleep, hives, use of medication (meds) to treat symptoms (sx), and use of medication to prevent symptoms) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4-days after each dose
Population: The safety population included all subjects who received at least 1 dose of vaccine, (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC + P80 Toddler Dose: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
- 13vPnC - P80 Toddler Dose: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
Arm/Group | 13vPnC + P80 Dose 1 Infant Series | 13vPnC - P 80 Dose 1 Infant Series | 13vPnC + P80 Dose 2 Infant Series | 13vPnC - P80 Dose 2 Infant Series | 13vPnC + P80 Dose 3 Infant Series | 13vPnC - P80 Dose 3 Infant Series | 13vPnC + P80 Toddler Dose | 13vPnC - P80 Toddler Dose
Number analyzed (Participants) | 250 | 250 | 246 | 249 | 246 | 247 | 240 | 244
Percentage of Participants
  Fv ≥38°C, ≤39°C(n=236,235,224,229,208,218,170,172) | 14.0 | 16.2 | 18.3 | 17.0 | 19.7 | 20.6 | 22.9 | 18.0
  Fv >39°C, ≤40°C(n=235,233,221,221,203,211,162,164) | 0.4 | 0.4 | 0.9 | 0.5 | 1.0 | 0.9 | 2.5 | 1.8
  Fv >40°C (n=235,233,221,221,203,211,160,164) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Decr appetite (n=237,237,221,224,210,222,172,183) | 21.5 | 22.4 | 16.3 | 24.1 | 21.4 | 20.7 | 26.2 | 29.0
  Irritability (n=240,239,232,232,215,226,184,198) | 55.0 | 55.2 | 51.7 | 53.9 | 45.6 | 50.0 | 49.5 | 56.1
  Incr sleep (n=242,242,231,229,209,221,174,182) | 46.3 | 52.5 | 35.9 | 39.3 | 25.8 | 27.6 | 19.0 | 30.8
  Decr sleep (n=238,236,227,227,209,217,170,180) | 35.7 | 29.7 | 24.7 | 26.4 | 25.4 | 24.4 | 19.4 | 25.6
  Meds-treat sx (n=236,235,222,226,205,218,172,168) | 14.0 | 16.6 | 15.3 | 16.8 | 15.1 | 14.7 | 21.5 | 15.5
  Meds-prevent sx(n=235,234,220,223,205,217,171,171) | 14.5 | 15.8 | 16.4 | 15.2 | 15.1 | 10.6 | 18.7 | 15.2

5. Primary Outcome: Geometric Mean Antibody Concentration (GMC) in 13vPnC+P80 Group Relative to 13vPnC-P80 Group After the 3-Dose Infant Series
Description: GMC as measured by enzyme-linked immunosorbent assay (ELISA) for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: One month after 3-dose infant series (at 5 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations, (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC + Polysorbate 80 After the Infant Series | 13vPnC - Polysorbate 80 After the Infant Series
Number analyzed (Participants) | 238 | 238
μg/mL
  Common Serotypes - Serotype 4 | 1.47 [1.30 to 1.65] | 1.53 [1.36 to 1.72]
  Common Serotypes - Serotype 6B | 0.51 [0.44 to 0.60] | 0.57 [0.48 to 0.68]
  Common Serotypes - Serotype 9V | 1.46 [1.34 to 1.60] | 1.51 [1.38 to 1.65]
  Common Serotypes - Serotype 14 | 2.37 [2.06 to 2.73] | 2.48 [2.20 to 2.80]
  Common Serotypes - Serotype 18C | 1.84 [1.67 to 2.03] | 1.87 [1.71 to 2.04]
  Common Serotypes - Serotype 19F | 1.46 [1.30 to 1.65] | 1.75 [1.60 to 1.91]
  Common Serotypes - Serotype 23F | 0.93 [0.83 to 1.05] | 1.11 [1.00 to 1.24]
  Additional Serotypes - Serotype 1 | 1.39 [1.26 to 1.55] | 1.48 [1.32 to 1.66]
  Additional Serotypes - Serotype 3 | 1.50 [1.38 to 1.63] | 1.62 [1.49 to 1.75]
  Additional Serotypes - Serotype 5 | 1.26 [1.13 to 1.40] | 1.30 [1.16 to 1.44]
  Additional Serotypes - Serotype 6A | 0.99 [0.88 to 1.12] | 1.04 [0.92 to 1.17]
  Additional Serotypes - Serotype 7F | 1.98 [1.81 to 2.15] | 1.89 [1.73 to 2.06]
  Additional Serotypes - Serotype 19A | 2.68 [2.44 to 2.95] | 2.94 [2.69 to 3.21]
Statistical Analysis 1: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 4 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for each common serotype was declared if the lower limit of the 2-sided 95% CI for the GMC ratio (13vPnC/7vPnC) > 0.5 (2-fold criterion); Difference = 0.96, 95% CI [0.81 to 1.13]
Statistical Analysis 2: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 6B the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.90, 95% CI [0.72 to 1.14]
Statistical Analysis 3: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 9V the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.97, 95% CI [0.85 to 1.10]
Statistical Analysis 4: Comparison: 13vPnC + Polysorbate 80 After the Infant Series; For serotype 14 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.96, 95% CI [0.79 to 1.15]
Statistical Analysis 5: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 18C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.98, 95% CI [0.86 to 1.13]
Statistical Analysis 6: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 19F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.84, 95% CI [0.72 to 0.97]
Statistical Analysis 7: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 23F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.84, 95% CI [0.71 to 0.98]
Statistical Analysis 8: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 1 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.94, 95% CI [0.81 to 1.10]
Statistical Analysis 9: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 3 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.93, 95% CI [0.83 to 1.04]
Statistical Analysis 10: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 5 the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.97, 95% CI [0.83 to 1.13]
Statistical Analysis 11: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 6A the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.96, 95% CI [0.81 to 1.13]
Statistical Analysis 12: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 7F the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 1.05, 95% CI [0.93 to 1.18]
Statistical Analysis 13: Comparison: 13vPnC + Polysorbate 80 After the Infant Series vs 13vPnC - Polysorbate 80 After the Infant Series; For serotype 19A the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Difference = 0.91, 95% CI [0.80 to 1.04]

6. Secondary Outcome: Geometric Mean Antibody Concentration (GMC) in 13vPnC Group Relative After the Toddler Dose
Description: as for outcome 5
Time Frame: one month after the toddler dose (at 13 months of age)
Population: Evaluable immunogenicity population had valid and determinate assay results, and had no other major protocol violations, (n) = number of participants with a determinate IgG antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC + Polysorbate 80 After Toddler Dose | 13vPnC - Polysorbate 80 After Toddler Dose
Number analyzed (Participants) | 227 | 238
μg/mL
  Common Serotypes - Serotype 4 (n=226,238) | 5.25 [4.65 to 5.92] | 5.38 [4.78 to 6.07]
  Common Serotypes - Serotype 6B (n=221,228) | 9.89 [8.70 to 11.23] | 10.65 [9.40 to 12.06]
  Common Serotypes - Serotype 9V (n=226,238) | 3.01 [2.73 to 3.31] | 3.10 [2.80 to 3.42]
  Common Serotypes - Serotype 14 (n=224,238) | 11.72 [10.26 to 13.40] | 11.95 [10.42 to 13.71]
  Common Serotypes - Serotype 18C (n=226,238) | 3.40 [3.06 to 3.78] | 3.10 [2.79 to 3.45]
  Common Serotypes - Serotype 19F (n=223,236) | 9.63 [8.45 to 10.97] | 10.27 [8.99 to 11.73]
  Common Serotypes - Serotype 23F (n=223,236) | 3.88 [3.44 to 4.38] | 4.15 [3.73 to 4.62]
  Additional Serotypes - Serotype 1 (n=226,238) | 6.03 [5.36 to 6.78] | 6.11 [5.43 to 6.87]
  Additional Serotypes - Serotype 3 (n=213,226) | 1.09 [0.99 to 1.20] | 1.16 [1.05 to 1.29]
  Additional Serotypes - Serotype 5 (n=225,234) | 3.80 [3.41 to 4.23] | 3.98 [3.59 to 4.41]
  Additional Serotypes - Serotype 6A (n=224,236) | 7.48 [6.66 to 8.40] | 8.19 [7.38 to 9.09]
  Additional Serotypes - Serotype 7F (n=226,238) | 5.36 [4.89 to 5.88] | 4.95 [4.50 to 5.44]
  Additional Serotypes - Serotype 19A (n=224,236) | 13.20 [11.88 to 14.67] | 13.02 [11.88 to 14.27]

ADVERSE EVENTS:
Groups:
- 13vPnC + P80 Infant Series; 13vPnC + P80 Post-Infant Series; 13vPnC + P80 Toddler Dose; 13vPnC + P80 6-Month Follow-up: Participants received one single 0.5mL dose of 13vPnC + P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
- 13vPnC - P 80 Infant Series; 13vPnC - P80 Post-Infant Series; 13vPnC - P80 Toddler Dose; 13vPnC - P80 6-Month Follow-up: Participants received one single 0.5mL dose of 13vPnC - P80 coadministered with Pentaxim and Engerix-B at 2 months of age, Pentaxim at 3 and 4 months age (infant doses), and Priorix at 12 months of age (toddler dose).
Arm/Group | 13vPnC + P80 Infant Series | 13vPnC - P 80 Infant Series | 13vPnC + P80 Post-Infant Series | 13vPnC - P80 Post-Infant Series | 13vPnC + P80 Toddler Dose | 13vPnC - P80 Toddler Dose | 13vPnC + P80 6-Month Follow-up | 13vPnC - P80 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 15/249 | 21/250 | 24/249 | 16/250 | 3/239 | 2/244 | 13/249 | 14/250
Other Adverse Events (participants affected / at risk) | 132/249 | 132/250 | 15/249 | 9/250 | 91/239 | 111/244 | 0/249 | 1/250
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC + P80 Infant Series (N=249) | 13vPnC - P 80 Infant Series (N=250) | 13vPnC + P80 Post-Infant Series (N=249) | 13vPnC - P80 Post-Infant Series (N=250) | 13vPnC + P80 Toddler Dose (N=239) | 13vPnC - P80 Toddler Dose (N=244) | 13vPnC + P80 6-Month Follow-up (N=249) | 13vPnC - P80 6-Month Follow-up (N=250)
Alloimmunisation (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath holding (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 9 | 5 | 1 | 0 | 1 | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 4 | 3 | 1 | 0 | 3 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fibrosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 4 | 3 | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Limbic traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meningitis meningococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 8 | 3 | 6 | 1 | 0 | 0 | 3 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal tubular disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ultrasound kidney abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC + P80 Infant Series (N=249) | 13vPnC - P 80 Infant Series (N=250) | 13vPnC + P80 Post-Infant Series (N=249) | 13vPnC - P80 Post-Infant Series (N=250) | 13vPnC + P80 Toddler Dose (N=239) | 13vPnC - P80 Toddler Dose (N=244) | 13vPnC + P80 6-Month Follow-up (N=249) | 13vPnC - P80 6-Month Follow-up (N=250)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Craniotabes (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brachycephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 5 | 2 | 1 | 0 | 0 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 11 | 0 | 0 | 4 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 4 | 0 | 0 | 1 | 1 | 0 | 0
Irritability (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 23 | 19 | 0 | 0 | 3 | 6 | 0 | 0
Rhinitis (Infections and infestations) | 19 | 21 | 3 | 1 | 8 | 10 | 0 | 0
Pharyngitis (Infections and infestations) | 17 | 15 | 0 | 0 | 10 | 19 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 17 | 13 | 0 | 0 | 9 | 17 | 0 | 0
Nasopharyngitis (Infections and infestations) | 13 | 13 | 1 | 0 | 4 | 10 | 0 | 0
Respiratory tract infection (Infections and infestations) | 8 | 6 | 0 | 0 | 2 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 0 | 0 | 3 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 4 | 0 | 0
Otitis media (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Exanthema subitum (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 5 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur functional (Investigations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased activity (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 14 | 7 | 3 | 1 | 2 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 8 | 1 | 2 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 45/181 | 59/181 | 0/0 | 0/0 | 75/178 | 81/188 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 43/176 | 63/176 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (any) (Skin and subcutaneous tissue disorders) | 41/167 | 38/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (any)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 4/179 | 8/178 | 0/0 | 0/0 | 4/160 | 2/165 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 1/172 | 1/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 2/163 | 2/165 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 39/179 | 55/183 | 0/0 | 0/0 | 52/174 | 63/181 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 46/178 | 62/175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Any)
Induration (Any) (Skin and subcutaneous tissue disorders) | 59/165 | 67/175 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (Any)
Induration (mild) (Skin and subcutaneous tissue disorders) | 33/179 | 41/180 | 0/0 | 0/0 | 45/169 | 53/178 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (mild) (Skin and subcutaneous tissue disorders) | 37/177 | 54/173 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild)
Induration (mild) (Skin and subcutaneous tissue disorders) | 51/165 | 56/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3;Induration (mild)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 18/179 | 28/182 | 0/0 | 0/0 | 20/164 | 34/171 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (moderate)=2.5 cm to 7.0 cm.
Induration (moderate) (Skin and subcutaneous tissue disorders) | 22/175 | 24/172 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (moderate) (Skin and subcutaneous tissue disorders) | 23/164 | 30/169 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/179 | 0/179 | 0/0 | 0/0 | 0/159 | 0/164 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/172 | 0/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/163 | 0/165 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 58/181 | 73/183 | 0/0 | 0/0 | 75/178 | 104/200 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (Any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 68/180 | 86/178 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Any)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 78/169 | 89/177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 56/181 | 63/180 | 0/0 | 0/0 | 63/176 | 90/194 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 centimeters (cm) to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 68/180 | 82/177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Mild)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 78/169 | 82/177 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 3/179 | 10/178 | 0/0 | 0/0 | 21/164 | 34/173 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 2/172 | 6/171 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Moderate)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 5/164 | 16/165 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/179 | 0/177 | 0/0 | 0/0 | 0/159 | 1/164 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/172 | 0/170 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (Severe)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/163 | 0/165 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (Severe)
Fever ≥38°C but ≤39°C (General disorders) | 33/236 | 38/235 | 0/0 | 0/0 | 39/170 | 31/172 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 41/224 | 39/229 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38°C but ≤39°C
Fever ≥38°C but ≤39°C (General disorders) | 41/208 | 45/218 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥38°C but ≤39°C
Fever >39°C but ≤40°C (General disorders) | 1/235 | 1/233 | 0/0 | 0/0 | 4/162 | 3/164 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 2/221 | 1/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39°C but ≤40°C
Fever >39°C but ≤40°C (General disorders) | 2/203 | 2/211 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >39°C but ≤40°C
Fever >40°C (General disorders) | 0/235 | 0/233 | 0/0 | 0/0 | 0/160 | 0/164 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40°C
Fever >40°C (General disorders) | 0/221 | 0/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40°C
Fever >40°C (General disorders) | 0/203 | 0/211 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever >40°C
Decreased appetite (General disorders) | 51/237 | 53/237 | 0/0 | 0/0 | 45/172 | 53/183 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 36/221 | 54/224 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 45/210 | 46/222 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Decreased sleep (General disorders) | 85/238 | 70/236 | 0/0 | 0/0 | 33/170 | 46/180 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 56/227 | 60/227 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 53/209 | 53/217 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep
Increased sleep (General disorders) | 112/242 | 127/242 | 0/0 | 0/0 | 33/174 | 56/182 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 83/231 | 90/229 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 54/209 | 61/221 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Irritability (General disorders) | 132/240 | 132/239 | 0/0 | 0/0 | 91/184 | 111/198 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 120/232 | 125/232 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 98/215 | 113/226 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.